CLINICAL TRIAL: NCT01359202
Title: "Spot Sign" Selection of Intracerebral Hemorrhage to Guide Hemostatic Therapy: SPOTLIGHT
Brief Title: "Spot Sign" Selection of Intracerebral Hemorrhage to Guide Hemostatic Therapy
Acronym: SPOTLIGHT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. David Gladstone (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Dr. David Gladstone, Principal Investigator - Sponsor, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Spotlight002
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Stroke
Keywords: Stroke; ICH; Intracerebral hemorrhage; acute stroke; rfVIIa; Niastase
MeSH Terms: conditions — Stroke; Cerebral Hemorrhage | interventions — recombinant FVIIa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Niastase RT (Active Comparator): Niastase RT 80ug/kg IV bolus
  Interventions: Biological: rfVIIa
- Placebo (Placebo Comparator): saline IV bolus
  Interventions: Other: Standard saline solution

INTERVENTIONS:
Biological: rfVIIa — 80ug/kg IV bolus
  Other Names: Niastase RT
  Arms: Niastase RT
Other: Standard saline solution — Saline
  Other Names: Saline solution sourced from local hospital
  Arms: Placebo

SUMMARY:
This clinical trial will enroll 110 patients from approximately 15 Canadian stroke centres. Patients coming to the emergency department with bleeding in the brain not due to trauma or other known causes who can be treated within 6 hours of onset will undergo CT angiography using standard CT scanners ("CAT scan"). Those with a "spot sign", a type of marker on the CT scan that shows the brain is still bleeding, will be randomly assigned to a single injection of "factor 7"(a blood clotting drug used in hemophilia) or placebo (inactive saline); patients without a spot sign will not be treated. The researchers will look at how much bleeding happens after the treatments are administered, as well as clinical outcomes such as death and disability. The researchers think that factor 7 will cause the bleeding to stop faster and possibly decrease death and disability.

DETAILED DESCRIPTION:
This phase II double blind RCT will enroll 110 patients from approximately 15 Canadian stroke centres. Acute ICH patients who can be treated within 6 hours of onset will undergo CT angiography using standard CT procedures. Those with a spot sign will be randomly assigned in a 1:1 ratio to a single injection of rFVIIa 80 µg/kg or placebo; patients without a spot sign will not be treated. The primary endpoint is ICH expansion within 24 hours.

ELIGIBILITY:
Inclusion Criteria

* Acute spontaneous primary supratentorial ICH diagnosed by CT scan.
* Presence of a spot sign within the hematoma on CTA source images
* Baseline ICH volume 3-90 ml
* Age 18 or older
* Investigator is able to randomize and administer study drug as soon as possible within a target of 60 minutes after CT angiogram and no later than 6 hours after stroke symptom onset (using the "last seen normal" principle).
* Plan to provide full medical care for at least 24 hours
* Assent-consent from patient or LAR prior to enrolment, or a waiver of consent (where REB approved) if patient/LAR assent-consent is not possible prior to enrolment.

Exclusion Criteria

* Brainstem or cerebellar hemorrhage.
* ICH secondary to known or suspected trauma, aneurysm, vascular malformation, hemorrhagic conversion of ischemic stroke, venous sinus thrombosis, thrombolytic treatment, tumour, or infection; or an in-hospital ICH or ICH as a result of any in-hospital procedure or illness.
* Baseline brain imaging shows evidence of acute or subacute ischemic stroke (chronic infarcts are not an exclusion).
* Contrast administration within the previous 24 hours.
* Evidence of thromboembolic risk factors, defined as any of the following: known history within the past 6 months of any of the following: (a) myocardial infarction, (b) coronary artery bypass surgery, (c) angina, (d) ischemic stroke, (e) transient ischemic attack, (f) carotid endarterectomy, (g) cerebral bypass surgery, (h) deep venous thrombosis, (i) pulmonary embolism, (j) any vascular angioplasty, stenting (coronary, peripheral vascular or cerebrovascular) or filter (e.g. vena cava filter);(k) prosthetic cardiac valve; and/or (l) known history of a high-risk thrombophilia (e.g. antithrombin III deficiency, antiphospholipid antibody syndrome, protein C deficiency, etc.)
* Known hereditary (e.g. hemophilia) or acquired hemorrhagic diathesis or coagulation factor deficiency.
* Any condition known that the investigator feels would pose a significant hazard if rFVIIa were administered.
* Planned surgery for ICH within 24 hours (placement of intraventricular catheter is not an exclusion).
* Planned withdrawal of care before 24 hours post-ICH onset.
* Known participation in another therapeutic trial.
* Known allergy or other contraindication to iodinated contrast dye.
* Known or suspected hypersensitivity to the trial product.
* Known unfractionated heparin use - must check PTT and exclude if elevated above upper limit of local lab's reference range.
* Known low-molecular weight heparin, heparinoid, factor X inhibitor, or direct thrombin inhibitor use within previous 7 days.
* Known GPIIb/IIIa antagonist use in previous 2 weeks.
* Known warfarin (or other anticoagulant) therapy with INR >1.40. Note: if the patient is suspected to have cirrhosis, study staff are to wait for the INR value prior to dosing, and ensure not to enroll the patient if the INR value is >1.40. Otherwise the physician should use their discretion if they believe the patient is not at risk for elevated INR.
* Concurrent or planned treatment with prothrombin complex concentrate, vitamin K, fresh frozen plasma, or platelet transfusion.
* Pregnancy or lactation. Women of childbearing potential must have a negative pregnancy test prior to randomization.
* Current clinical symptoms suggestive of acute coronary ischemia (e.g. chest pain).
* Baseline ECG evidence of acute coronary ischemia (e.g. ST elevation in 2 contiguous leads, new LBBB, ST depression).
* Baseline platelet count <50,000 or INR >1.40 or elevated PTT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
ICH size | 24 hours
  Difference between groups in ICH size on CT scan at 24 hours post-dose, adjusted for baseline ICH size

SECONDARY OUTCOMES:
Feasibility | 0
  Percentage of sites who can meet recruitment targets of 2 patients per site per year; % patients who meet the target time of <45 minutes from emergency department arrival to the start of the scan; % patients who meet the target time of <60 minutes from the end of the CT angiogram to administration of study drug; Local site spot sign interpretation accuracy as judged by central adjudicator; protocol violations
Waiver of consent process evaluation/effectiveness | 4,90 days
  Waiver of consent use, acceptability, and effect on treatment times. Questionnaire will be administed to subject/LAR at 4 days and 90 days.
Acute blood pressure control | 1hr
  % subjects where blood pressure control was acheived, defined as achieving systolic BP <180 mmHg within 1 hour post-randomization
Thromboembolic events | 4 days
  Incidence of myocardial infarction and ischemic stroke within 4 days; any other arterial or venous thromboembolic SAEs within 4 days
Mortality | 90 days
  90-day mortality rate
Unstable angina | 4 days
  Unstable angina w/in 4 days of treatment
Troponin increase | 4 days
  Troponin rise above upper limit of normal within 4 days (without clinical symptoms or ECG evidence of acute coronary syndrome)
DVT | 4 days
  Deep venous thrombosis (DVT) within 4 days
Pulmonary embolism | 30 days
  PE within 30 days
Cognition | 90 days, 1 year
  Montreal Cognitive Assessment (MoCA) and Stroke Impact Scale at 90 days and 1 year.
Disability | 90 d, 1 year
  Proportion of subjects with modified Rankin score 5-6 (death or severe disability) at 90 days and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David J Gladstone, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Richard Aviv, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Andrew Demchuk, MD, Principal Investigator — University of Calgary
Locations (15):
- Canada (15):
  - Foothills Medical Centre, Calgary, Alberta
  - Walter C. Mackenzie Health Sciences Centre, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Vancouver Island Health Authority, Victoria, British Columbia
  - Hamilton HSC, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Hôpital Charles Le Moyne, Greenfield Park, Quebec
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - Montreal Neurological Institute, Montreal, Quebec

REFERENCES:
- [Derived] Al-Ajlan FS, Gladstone DJ, Song D, Thorpe KE, Swartz RH, Butcher KS, Del Campo M, Dowlatshahi D, Gensicke H, Lee GJ, Flaherty ML, Hill MD, Aviv RI, Demchuk AM; SPOTLIGHT Investigators. Time Course of Early Hematoma Expansion in Acute Spot-Sign Positive Intracerebral Hemorrhage: Prespecified Analysis of the SPOTLIGHT Randomized Clinical Trial. Stroke. 2023 Mar;54(3):715-721. doi: 10.1161/STROKEAHA.121.038475. Epub 2023 Feb 9. PMID 36756899
- [Derived] Gladstone DJ, Aviv RI, Demchuk AM, Hill MD, Thorpe KE, Khoury JC, Sucharew HJ, Al-Ajlan F, Butcher K, Dowlatshahi D, Gubitz G, De Masi S, Hall J, Gregg D, Mamdani M, Shamy M, Swartz RH, Del Campo CM, Cucchiara B, Panagos P, Goldstein JN, Carrozzella J, Jauch EC, Broderick JP, Flaherty ML; SPOTLIGHT and STOP-IT Investigators and Coordinators. Effect of Recombinant Activated Coagulation Factor VII on Hemorrhage Expansion Among Patients With Spot Sign-Positive Acute Intracerebral Hemorrhage: The SPOTLIGHT and STOP-IT Randomized Clinical Trials. JAMA Neurol. 2019 Dec 1;76(12):1493-1501. doi: 10.1001/jamaneurol.2019.2636. PMID 31424491